CLINICAL TRIAL: NCT01331733
Title: Comparative Assessment of the Clinical Utility of Ovarian Stimulation With Menotropin Versus Menotropin Plus GnRH Antagonist Following Two Protocols of Ovulation Induction for Intrauterine Insemination
Brief Title: Comparative Assessment of the Clinical Utility of Ovarian Stimulation With Menotropin Versus Menotropin Plus GnRH Antagonist
Acronym: PROMENIA
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring SAU (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Other Study IDs: FER-MEN-2006-01
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Sterility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hMG-HP: Patients with a condition
  Interventions: Drug: hMG-HP
- hMG-HP + GnRH antagonist: Patients with a condition
  Interventions: Drug: hMG + GnRH antagonist

INTERVENTIONS:
Drug: hMG-HP
  Groups: hMG-HP
Drug: hMG + GnRH antagonist
  Groups: hMG-HP + GnRH antagonist

SUMMARY:
To assess the effectiveness of protocols of ovarian hyperstimulation combining urinary gonadotrophins + GnRH antagonist vs urinary gonadotrophins, to achieve clinical pregnancy in females undergoing intrauterine insemination.

Study hypothesis: protocols combining urinary gonadotrophins + GnRH antagonist should be more effective than monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-36 years
* Body mass index (BMI) between 18 and 26
* Prolactin within the laboratory normal range
* Couples affected by sterility able to treat by IUI (intrauterine insemination)
* Patients undergoing Menopur® treatment
* Normal thyroid function
* Regular menses (21-35 days)
* Couples willing to participate in the study that have signed the informed consent form
* Seminal sample REM>3 million

Exclusion Criteria:

* Two previous ART (assisted reproductive technology) cycles without ongoing pregnancy
* Policystic ovarian syndrome
* Evidence of significant bacterial infection in the seminogram of the couple in the preceding 6 months

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females affected by sterility able to undergo intrauterine insemination
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 30 days

SECONDARY OUTCOMES:
Live birth rate | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (7):
- Spain (7):
  - Investigational site, Barcelona, Barcelona
  - Investigational site, Ciudad Real, Ciudad Real
  - Investigational site, Girona, Gerona
  - Investigational site, La Rioja, La Rioja
  - Investigational site, Navarra, Navarre
  - Investigational site, Reus, Tarragona
  - Investigational site, Valladolid, Valladolid